CLINICAL TRIAL: NCT04047329
Title: Risk Factors and Impact of Anesthesia Techniques on Myocardial Infarction Following Transurethral Resection of the Prostate: a Nationwide Database Case Control Study
Brief Title: Risk Factors and Impact of Anesthesia Techniques on Myocardial Infarction Following Transurethral Resection of the Prostate
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 104-6697B
Record Dates: First submitted 2019-07-23; First posted 2019-08-06 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2015-09

CONDITIONS: Anesthesia; Transurethral Resection of Prostate Syndrome; Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Anesthesia, General

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Without post-operative myocardial infarction: Patients without post-operative myocardial infarction after first admission for transurethral resection of the prostate
  Interventions: Other: general anesthesia or neuraxial anesthesia
- With post-operative myocardial infarction: Patients with post-operative myocardial infarction after first admission for transurethral resection of the prostate
  Interventions: Other: general anesthesia or neuraxial anesthesia

INTERVENTIONS:
Other: general anesthesia or neuraxial anesthesia

SUMMARY:
This study examined the risk factors and the influence of the type of anesthetic used during transurethral resection of the prostate (TURP) on subsequent incidence of myocardial infarction (MI).

DETAILED DESCRIPTION:
This study utilized a population-based, nationwide dataset to evaluate the risk factors of MI for patients with benign prostate hypertrophy (BPH) who received TURP. Besides, The study also compared the different effects of general anesthesia (GA) and neuraxial anesthesia (NA) on the incidence of MI within 6 and 12 months after TURP.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving TURP surgery (1998-2012)

Exclusion Criteria:

* Patients without anesthesia records
* Patients receiving both general and neuraxial anesthesia
* Mortality within 12 months of TURP

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving TURP
Sampling Method: Non-Probability Sample
Enrollment: 115025 (Actual)
Dates: Start 1998-01-01 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2016-03-22 (Actual)

PRIMARY OUTCOMES:
Postoperative myocardial infarction | within 6 months after the first admission for TURP
  Patients experienced myocardial infarction after transurethral resection of the prostate (TURP)
Postoperative myocardial infarction | within 12 months after the first admission for TURP
  Patients experienced myocardial infarction after transurethral resection of the prostate (TURP)
Patient's age (year-old) that developed post-TURP myocardial infarction | within 6 months after the first admission for TURP
  We analyze age distribution of patients with post-TURP myocardial infarction
Patient's age (year-old) that developed post-TURP myocardial infarction | within 12 months after the first admission for TURP
  We analyze age distribution of patients with post-TURP myocardial infarction
Number of patients with pre-operative diagnosed Diabetes Mellitus developing post-TURP myocardial infarction | within 6 months after the first admission for TURP
  We analyze pre-operative diagnosed Diabetes Mellitus rate in patients who had myocardial infarction after the surgery of TURP.
Number of patients with pre-operative diagnosed Diabetes Mellitus developing post-TURP myocardial infarction | within 12 months after the first admission for TURP
  We analyze pre-operative diagnosed Diabetes Mellitus rate in patients who had myocardial infarction after the surgery of TURP.
Number of patients with pre-operative diagnosed disorders of lipoid metabolism developing post-TURP myocardial infarction | within 6 months after the first admission for TURP
  We analyze pre-operative diagnosed disorders of lipoid metabolism rate in patients who had myocardial infarction after the surgery of TURP.
Number of patients with pre-operative diagnosed disorders of lipoid metabolism developing post-TURP myocardial infarction | within 12 months after the first admission for TURP
  We analyze pre-operative diagnosed disorders of lipoid metabolism rate in patients who had myocardial infarction after the surgery of TURP.
Number of patients with pre-operative diagnosed gout developing post-TURP myocardial infarction | within 6 months after the first admission for TURP
  We analyze pre-operative diagnosed gout rate in patients who had myocardial infarction after the surgery of TURP.
Number of patients with pre-operative diagnosed gout developing post-TURP myocardial infarction | within 12 months after the first admission for TURP
  We analyze pre-operative diagnosed gout rate in patients who had myocardial infarction after the surgery of TURP.
Number of patients with pre-operative diagnosed hypertension developing post-TURP myocardial infarction | within 6 months after the first admission for TURP
  We analyze pre-operative diagnosed hypertension rate in patients who had myocardial infarction after the surgery of TURP.
Number of patients with pre-operative diagnosed hypertension developing post-TURP myocardial infarction | within 12 months after the first admission for TURP
  We analyze pre-operative diagnosed hypertension rate in patients who had myocardial infarction after the surgery of TURP.
Number of patients with pre-operative diagnosed heart disease history developing post-TURP myocardial infarction | within 6 months after the first admission for TURP
  We analyze pre-operative diagnosed heart disease rate in patients who had myocardial infarction after the surgery of TURP.
Number of patients with pre-operative diagnosed heart disease history developing post-TURP myocardial infarction | within 12 months after the first admission for TURP
  We analyze pre-operative diagnosed heart disease rate in patients who had myocardial infarction after the surgery of TURP.
Number of patients with pre-operative diagnosed stroke history developing post-TURP myocardial infarction | within 6 months after the first admission for TURP
  We analyze pre-operative diagnosed stroke rate in patients who had myocardial infarction after the surgery of TURP.
Number of patients with pre-operative diagnosed stroke history developing post-TURP myocardial infarction | within 12 months after the first admission for TURP
  We analyze pre-operative diagnosed stroke rate in patients who had myocardial infarction after the surgery of TURP.
Number of patients with pre-operative diagnosed liver cirrhosis history developing post-TURP myocardial infarction | within 6 months after the first admission for TURP
  We analyze pre-operative diagnosed liver cirrhosis rate in patients who had myocardial infarction after the surgery of TURP.
Number of patients with pre-operative diagnosed liver cirrhosis history developing post-TURP myocardial infarction | within 12 months after the first admission for TURP
  We analyze pre-operative diagnosed liver cirrhosis rate in patients who had myocardial infarction after the surgery of TURP.
Number of patients with pre-operative diagnosed chronic obstructive pulmonary disease developing post-TURP myocardial infarction | within 6 months after the first admission for TURP
  We analyze pre-operative diagnosed chronic obstructive pulmonary disease rate in patients who had myocardial infarction after the surgery of TURP.
Number of patients with pre-operative diagnosed chronic obstructive pulmonary disease developing post-TURP myocardial infarction | within 12 months after the first admission for TURP
  We analyze pre-operative diagnosed chronic obstructive pulmonary disease rate in patients who had myocardial infarction after the surgery of TURP.
Number of patients with pre-operative diagnosed asthma developing post-TURP myocardial infarction | within 6 months after the first admission for TURP
  We analyze pre-operative diagnosed asthma rate in patients who had myocardial infarction after the surgery of TURP.
Number of patients with pre-operative diagnosed asthma developing post-TURP myocardial infarction | within 12 months after the first admission for TURP
  We analyze pre-operative diagnosed asthma rate in patients who had myocardial infarction after the surgery of TURP.

SECONDARY OUTCOMES:
Number of patients who had post-operative myocardial infarction after receiving general anesthesia for TURP | within 6 months after the first admission for TURP
  Number of patients who had post-operative myocardial infarction after receiving general anesthesia for TURP
Number of patients who had post-operative myocardial infarction after receiving neuraxial anesthesia for TURP | within 6 months after the first admission for TURP
  Number of patients who had post-operative myocardial infarction after receiving neuraxial anesthesia for TURP
Number of patients who did not have post-operative myocardial infarction after receiving general anesthesia for TURP | within 12 months after the first admission for TURP
  Number of patients who did not have post-operative myocardial infarction after receiving general anesthesia for TURP
Number of patients who did not have post-operative myocardial infarction after receiving neuraxial anesthesia for TURP | within 12 months after the first admission for TURP
  Number of patients who did not have post-operative myocardial infarction after receiving neuraxial anesthesia for TURP